CLINICAL TRIAL: NCT06891820
Title: Multifaceted Analysis of the Adaptation of Rowers in the Process of Sports Training
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Rowers 2025
Record Dates: First submitted 2025-03-03; First posted 2025-03-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-02

CONDITIONS: Ferroptosis; Inflammation; Muscle Damage; Nervous System Diseases
MeSH Terms: conditions — Inflammation; Nervous System Diseases | interventions — Physical Exertion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Polyethylene tubes (4.9 ml) containing dipotassium ethylenediaminetetraacetic acid (EDTAK2) anticoagulant.
  2. Polyethylene clotting activator tubes (9 ml)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Physical effort: Rowers will perform an intensive exercise test on a rowing ergometer (Concept II, USA), covering a distance of 2000 meters in the shortest time possible. The test on the rowing ergometer will be performed under the supervision of a physician.
  Interventions: Other: Physical effort

INTERVENTIONS:
Other: Physical effort — The examined athletes will be subjected to an effort on a rowing ergometer, covering a designated distance in the shortest possible time.

SUMMARY:
This study aims to analyze in detail selected indicators of appetite regulation, metabolism, and iron balance in competitive rowers undergoing intense exercise. The project involves assessing dynamic hormonal and biochemical changes in the athletes' bodies, which will allow a better understanding of the body's adaptive mechanisms to prolonged physical strain.

Research group: the research will be conducted in a homogeneous group of professional rowers (N=30), all competitors qualified for the Polish Youth Rowing Team:

* aged 19 - 24, because the age group must be homogeneous,
* the size of the group is about thirty people, which in the case of a homogeneous group will enable statistical analyzes to be conducted.

Rowing performance test: At the beginning and end of the training camp, participants will perform a test on a rowing ergometer (Concept II, USA). Each subject will have to cover a distance of 2000 m in the shortest possible time, which is the distance starting in rowing competitions. The results of both tests will be considered in the selection for the championship team; therefore, athletes will be well motivated to perform both tests with maximum effort.

Blood samples will be taken from the cubital vein at three-time points: before each ergometer test (after overnight fasting), directly after the test, and after a 1-hour recovery period.

DETAILED DESCRIPTION:
The study aims to conduct a detailed analysis of selected indicators of appetite regulation, metabolism, inflammation, and iron balance in competitive rowers undergoing intense exercise. The project involves assessing dynamic hormonal and biochemical changes in the athletes' bodies, which will allow for a better understanding of the body's adaptive mechanisms to prolonged physical strain.

Research group: The research will be conducted in a homogeneous group of professional rowers (N=30), all competitors qualified for the Polish Youth. Rowing Team:

* aged 19 - 24, because the age group must be homogeneous,
* the size of the group is about thirty people, which in the case of a homogeneous group will enable statistical analyzes to be conducted.

Rowing performance test: at the beginning and at the end of the training camp, participants will perform a test on a rowing ergometer (Concept II, USA), each subject will have to cover a distance of 2000 m in the shortest possible time, which is the distance starting in rowing competitions. The results of both tests will be considered in the selection for the championship team; therefore, athletes will be well motivated to perform both tests with maximum effort.

Blood samples will be taken from the cubital vein at three-time points: before each ergometer test (after overnight fasting), directly after the test, and after a 1-hour recovery period.

Measurement: All determined parameters will be measured with the available equipment in the biochemical laboratory of Poznan University of Physical Education, Faculty of Sport Sciences in Gorzow Wlkp., using commercial assay kits. Measurements will be performed by the project contractors.

1. Polyethylene tubes (4.9 ml) containing dipotassium ethylenediaminetetraacetic acid (EDTAK2) anticoagulant will be used for the following tests:

   (a) complete blood count (18 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). White blood cell indices: WBC (white blood cells), LYM (lymphocytes as a percentage), LYM (lymphocytes), MON (monocytes as a percentage), MON (monocytes), GRA (granulocytes as a percentage), GRA (granulocytes). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood cells Distribution Width). Platelet indices: PLT (Platelet), MPV (Mean Platelet Volume), PDW (Platelet Distribution Width), PCT (Thrombocrit) (b) gene expression.
2. Polyethylene clotting activator tubes (9 ml) will be centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum will be pipetted into several Eppendorf tubes, which will then be frozen (temp. -80°C). All the following biochemical parameters will be determined from the extracted serum: using the ELISA method by the test manufacturer's instructions. The designations include the flowing parameters:

   1. Analysis of leptin, ghrelin, glucagon-like peptide-1 (GLP-1), peptide YY (PYY), pancreatic polypeptide (PP) and cholecystokinin (CCK) levels will allow assessment of dynamic hormonal changes in rowers in relation to training intensity, energy availability and diet composition.

      * Leptin (LEP) - a satiety hormone whose levels may be reduced in athletes with low levels of body fat.
      * Ghrelin (GHRL) - a hunger hormone that increases in states of energy deficit and may affect the regulation of caloric intake.
      * GLP-1, PYY, PP and CCK - intestinal peptides involved in appetite suppression and modulation of insulin secretion and fat metabolism.
   2. Biochemical and hormonal parameters

      Stress and recovery hormones:
      * Cortisol - a marker of stress response and catabolism.
      * Testosterone - a key anabolic hormone, whose ratio to cortisol (T/C) helps assess the balance between anabolism and catabolism.

      Neurotransmitters associated with fatigue resistance:
      * Serotonin - important in regulating mood and central fatigue; its excess can contribute to lethargy and decreased motivation.
      * Dopamine - crucial for motivation and mental performance; decreased levels may indicate neurotransmitter depletion.

      Sex hormones and metabolic balance:
      * Estradiol
      * Progesterone - in women indicators of menstrual cycle and hormonal balance,
   3. ferroptosis parameters

      * antioxidants: glutathione (GSH), glutathione peroxidase 4 (GPX4),
      * markers of oxidative stress: 4-Hydroxynonenal (4-HNE), Heme oxygenase 1 (HO-1)
      * iron status parameters: soluble transferrin receptor, ferritin, erythroferrone, lactoferrin

      The iron and Total Iron Binding Capacity (TIBC) levels will be determined using the colorimetric method on the SPECTROstar Nano reader. Unsaturated Iron Binding Capacity (UIBC) will be calculated from the formula: UIBC = TIBC-iron in serum)
   4. Markers of energy metabolism:

      * Glucose - a key energy source for working muscles, to assess how the body regulates carbohydrate metabolism during and after exercise.
      * Glycogen - an important indicator of energy reserve utilization during high intensities, to determine the level of energy reserve utilization.
      * Insulin - responsible for the transport of glucose into muscle cells and to assess how the body manages energy before, during and after exercise, and whether adaptation to load is effective,
      * Lactic acid - an indicator of exercise intensity and the balance between aerobic and anaerobic metabolism.

   Markers of muscle damage:
   * CK (creatine kinase), myoglobin - increases with muscle damage, especially after intense exercise, allows to assess the degree of fatigue and risk of overtraining.
   * interleukin-6 (IL-6) - mediator of inflammatory response and marker of fatigue; rises after intense exercise, indicates fatigue and recovery processes.

   Markers of metabolic adaptation and recovery:

   - fibroblast growth factor-21 (FGF-21) - , a protein, regulates metabolism and restoration of energy resources, allows assessment of the body's adaptation to intense exercise.
3. Using a portable analyzer system for measuring blood gas, electrolytes and metabolites (epoc®), using dedicated epoc® test cards. Measured parameters: Direct: pH, partial pressure of carbon dioxide (pCO2), partial pressure of oxygen (pO2), total plasma carbon dioxide (tCO2), sodium (Na+), potassium (K+), calcium (Ca++), chlorine (Cl-), hematocrit (Hct), glukose (glu), Lactic Acid (Lac), Crea, Urea, urea nitrogen (BUN). Calculated values: cHgb, bicarbonate level (cHCO3), cTCO2, excess base in extracellular fluid (BE ecf), BE(b), total blood saturation (cSO2), glomerular filtration rate (GFRmdr), GFRmdr-a, GFRckd, GFRckd-a, GFRswz, anion gap (AGAP), AGapK, BUN/Crea, Urea/Crea. It will be determined from capillary blood taken from the earlobe (90 µl). Lactic acid will be determined from capillary blood taken from the earlobe (10 µl). The determination will be performed with dedicated reagents, using a portable biochemical photometer Vario Photometer II (Diaglobal, Berlin, Germany).

ELIGIBILITY:
1. Inclusion Criteria:

   * consent to participate in the study,
   * regular training regimen,
   * current medical examination,
   * no health contraindications (to be decided by a doctor).
2. Exclusion Criteria:

   * Lack of consent for blood draws,
   * injuries,
   * health problems,
   * anti-inflammatory drugs,
   * supportive substances, supplements in the last 3 months before the start of the study.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Polish Youth Rowing Team
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
The Blood morphology | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Using MYTHIC18 hematology analyzer (Cormay Diagnostics, Geneva, Switzerland). Qualitative and quantitative evaluation of morphological elements of blood (determination in venous blood).
Changes from baseline in Glycogen level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of glycogen [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline Insulin level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of insulin [μIU/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baselineCreatine kinase activity (CK) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concetration of CK [ng/ml]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline interleukin-6 (Il-6) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Il-6 [pg/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in fibroblast growth factor 21 (FGF-21) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of FGF-21 [pg/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in lactic acid (LA) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concetration of LA [mmol/l]. Using a portable biochemical photometer Vario Photometer II (Diaglobal, Berlin, Germany) (capillary blood from the ear lobe).
Gene expression | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Genes studied: LEP, GHRL, AGRP, GOT1 and GPX4.
  RNA isolation will be performed by the column method on the Direct-zol™ RNA MiniPrep Plus Kits, according to the test manufacturer's instructions. Gene expression analysis from cells isolated from blood will be performed by reverse transcription using TaqMan
Changes from baseline in testosterone level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of testosterone [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in serotonin level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery
  Concentration of serotonin [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in progesterone level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery
  Concentration of progesterone [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in estradiol level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery
  Concentration of estradiol [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in dopamine level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery
  Concentration of dopamine [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Baseline Mood Profile of Athletes Before Exercise Test Using POMS Questionnaire. | At rest (before the exercise test).
  The Profile of Mood States (POMS) questionnaire measures mood states and emotional well-being.
Baseline Mental Toughness in Sport measured using the Scale of Mental Toughness in Sport (SMTQ) | At rest (before the exercise test).
  Scale of Mental Toughness in Sport (SMTQ) - to assess an athlete's ability to cope with training loads and stress
Baseline Eating Behavior and Attitudes of Athletes Before Exercise Test Using EDE-Q 6.0 Questionnaire. | At rest (before the exercise test).
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder behaviors and attitudes.
Baseline Appetite Assessment of Athletes Before Exercise Test Using Visual Analogue Scale (VAS). | At rest (before the exercise test).
  The Visual Analogue Scale (VAS) measures subjective appetite sensations-linear scale from one to 10 where 10 is the strongest feeling.
Changes from baseline in leptin(LEP) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Satiety regulation marker. Concentration of leptin [pg/ml].ELISA method by the test manufacturer's instructions.
Changes from baseline in glucagon-like peptide-1 (GLP-1) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Satiety regulation marker. Concentration of GLP-1 [pg/ml]. ELISA method by the test manufacturer's instructions.
Changes from baseline in peptide YY (PYY) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Satiety regulation marker. Concentration of leptin [pg/ml]. ELISA method by the test manufacturer's instructions.
Changes from baseline in pancreatic polipeptide (PP) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Satiety regulation marker. Concentration of PP [pg/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in ghrelin (GHRL) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Hunger regulation marker. Concentration of GHRL [pg/ml].ELISA method by the test manufacturer's instructions.
Changes from baseline in cholocystokinin (CCK) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Satiety regulation marker. Concentration of CCK [pg/ml].ELISA method by the test manufacturer's instructions.
Changes from baseline in Soluble transferrin receptor level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Soluble transferrin receptor [μg/ml]. ELISA method by the test manufacturer's instructions.
Changes from baseline in Ferritin level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of ferritin [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in 4-Hydroxynonenal (4-HNE) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of 4-Hydroxynonenal (4-HNE) [pg/ml]. ELISA method by the test manufacturer's instructions
Changes from baseline in Glutathione Peroxidase 4 (GPX4) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Human Glutathione Peroxidase 4 (GPX4) [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Glutathione level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Glutathione (GSH) [μg/mL]. ELISA method by the test manufacturer's instructions.
Changes from baseline in Heme Oxygenase 1(HO-1) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Heme Oxygenase 1 (HO-1) [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Erythroferrone level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of erythroferrone [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Lactoferrin level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of lactoferrin [ng/mL]. ELISA method by the test manufacturer's instructions
Changes from baseline in Iron (Fe) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  The iron level [µg/dL] will be determined using the colorimetric method on the SPECTROstar Nano reader.
Changes from baseline in acid-base balance - urea nitrogen (BUN) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of BUN [ml/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - anion gap (AGAP) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of AGAP [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - excess base in extracellular fluid (BE ecf) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Be ecf [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - sodium (Na) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Na [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - calcium (Ca) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Ca [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - potassium (K) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of K [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - chlorine (Cl) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of Cl [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - bicarbonate level (cHCO3). | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of cHCO3 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - total plasma CO2 (tCO2) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of tCO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - partial pressure of carbon dioxide (pCO2) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of pCO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - partial pressure of oxygen (pO2) | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of pO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance -total blood saturation (cSO2) level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of cSO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - urea level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of urea [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - crea level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of crea [mg/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - hematocrit [hct] level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of hct [%]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - hemoglobin [chgb] level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of chgb [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - glukose [glu] level. | At rest (before the test), directly after the test, and after a 1-hour recovery period.
  Concentration of glu [mg/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).

SECONDARY OUTCOMES:
Antropometric characteristic - height | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Antropometric characteristic - weight | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including weight (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Antropometric characteristic - LBM | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including lean body mas (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Antropometric characteristic - TBW | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including total body water (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Antropometric characteristic - Water% | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including water (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [%]
Antropometric characteristic - FAT | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including fat (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [%]
Food record - energy | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: energy [kcal]
Food record - protein | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: protein [g]
Food record - carobhydrates | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: carbohydrates [g]
Food record - fiber | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fiber [g]
Food record - fat | Day before the Day 1, in the morning at Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fat [g]

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejborn, Professor, Study Director — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No